CLINICAL TRIAL: NCT06425068
Title: Assessment of an Innovative Air Mattress on Critically Ill Infants
Acronym: Prepicare
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Simon Annaheim (Other)
Collaborators: University Children's Hospital, Zurich (Other)
Responsible Party: Sponsor-Investigator, Simon Annaheim, Principle Investigator, Empa, Swiss Federal Laboratories for Materials Science and Technology
Organization: Empa, Swiss Federal Laboratories for Materials Science and Technology (Other)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: Empa PSP 5211.02071
Record Dates: First submitted 2024-04-11; First posted 2024-05-22 (Actual); Last update posted 2025-01-13 (Actual); Status verified 2025-01

CONDITIONS: Skin Abnormalities; Skin; Injury, Superficial; Skin; Ulcer, Decubitus
Keywords: Air mattress; Skin interface pressure; Skin contact area; Lying comfort
MeSH Terms: conditions — Skin Abnormalities; Wounds and Injuries; Pressure Ulcer

STUDY DESIGN:
Intervention Model Description: The study population comprises 26 patients being exposed to the conventional foam mattress (active comparator) and the novel air mattress (experimental) for one hour each in a random order. Interface pressure and contact are will be measured by means of a pressure mattress applied on top of the support systems. The patient comfort will be assessed objectively based on vital sign readings and subjectively based on questionnaire filled by professional care personnel and parents.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Investigation of contact pressure distribution in a novel air mattress (Experimental): Exposure of the patient to the novel air mattress. Recording of interface pressure and contact area between the patient and the air mattress for one hour.
  Regular measurement of vital signs and comfort and assessment of risk to develop side effects, particularly skin pressure injuries.
  Interventions: Device: Exposure of the patient to a novel air mattress.
- Investigation of contact pressure distribution in a conventional foam mattress (Active Comparator): Exposure of the patient to the conventional foam mattress. Recording of interface pressure and contact area between the patient and the foam mattress for one hour.
  Regular measurement of vital signs and comfort and assessment of risk to develop side effects, particularly skin pressure injuries.
  Interventions: Device: Exposure of the patient to a conventional foam mattress.

INTERVENTIONS:
Device: Exposure of the patient to a novel air mattress. — see information provided in the "Arms" section (experimental)
  Arms: Investigation of contact pressure distribution in a novel air mattress
Device: Exposure of the patient to a conventional foam mattress. — see information provided in the "Arms" section (active comparator)
  Arms: Investigation of contact pressure distribution in a conventional foam mattress

SUMMARY:
The permanent bedding of critically ill neonates and infants in the pediatric intensive care unit (PICU) for an extended amount of time can result in the development of pressure injuries (PI). PIs can form due to high and permanent local interface pressure induced by contact with bed surfaces or other medical devices. The currently used state-of-the-art support systems consist of conventional foam mattresses. In this study, the investigators explore the effect of a newly developed air mattress with regard to contact are and reduction in the average interface pressure in infants assigned to the pediatric intensive care unit of the childrens hospital in Zurich.

DETAILED DESCRIPTION:
The permanent bedding of critically ill neonates and infants in the pediatric intensive care unit (PICU) for an extended amount of time can result in the development of pressure injuries (PI). This results in a further prolongation of the hospital stay, additional suffering of the patient, scarring, increased mortality and morbidity, and increased healthcare costs. Infants are at particular risk since their skin hasn't matured yet and is mechanically weak, and for example neonates lack a robust stratum corneum entirely. Furthermore, the thickness of their skin is reduced by 60% when compared to skin of adults. Thus, pressure cannot be equally absorbed leading to higher tissue internal stress. PIs can form due to high and permanent local interface pressure induced by contact with bed surfaces or other medical devices. Contact pressure can hamper blood flow in subcutaneous areas, increasing susceptibility for pressure injuries. While sophisticated equipment to manage the interface pressure and reduce the risk of developing pressure injuries is abundant for adults, very little is designed explicitly for neonates and infants. The currently available air mattresses are not being used due to safety concerns and impracticability. Furthermore, they are designed for infants from half a year of age and, thus, not considering the low body weight of premature babies or neonates. This is why the currently used conventional foam mattresses remain first choice. However, foam mattresses are designed for optimal support of a specific weight and, therefore, making them unsuitable for the use as a one-fits-all solution in a highly heterogenic patient cohort. In addition, compressed foam gets stiffer at compressed areas, increasing the local pressure impact and, thus, PI risk. On the other hand, the structures of the hereby-developed air mattress can freely move and optimally adjust to the patient's body shape. This increases contact area, reduces the average interface pressure and blunts local pressure peaks at the areas with the most indentation, ensuring a more homogenous pressure distribution at a lower level. This ultimately is expected to result in a lower PI incidence. As a side effect, lying comfort for the patient will be increased.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent signed by the legal guardian
* Admitted to the pediatric intensive care unit (PICU)
* Age: late preterm (>34 gestational age) up to 6 months
* Admission at least 24 hours to PICU prior to intervention
* Presence/availability of at least one parent/legal guardian

Exclusion Criteria:

* Life threatening condition
* Patients who cannot be positioned in supine position
* Skin injury at body area in contact with support surface
* Patients with congenital skin disorders
* Patients with omphalocele or gastroschisis
* Newborns with peripartum asphyxia and hypothermia therapy
* Language communication difficulties with the legal guardians
* Surgical patients on the day of surgery
* birth weight <1250g

Ages: 10 Days to 6 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 23 (Actual)
Dates: Start 2024-05-07 (Actual); Primary Completion 2024-09-10 (Actual); Study Completion 2024-09-10 (Actual)

PRIMARY OUTCOMES:
Interface pressure resulting from the exposure of patients to the supportive structures as measured by a pressure sensitive mat (xsensor, LX100:100.160.05, XSENSOR Technology Corporation, Calgary, Canada). | baseline
  Quantification of interface pressure between the patient and the mattress surfaces with emphasis on data of highest pressures (median for top 25% of pressure data observed; 4th quartile of pressure data).
Interface pressure resulting from the exposure of patients to the supportive structures as measured by a pressure sensitive mat (xsensor, LX100:100.160.05, XSENSOR Technology Corporation, Calgary, Canada). | after 60 minutes of exposure to the mattress
  Quantification of interface pressure between the patient and the mattress surfaces with emphasis on data of highest pressures (median for top 25% of pressure data observed; 4th quartile of pressure data).

SECONDARY OUTCOMES:
Contact area resulting from the exposure of patients to the supportive structures as detected by a pressure sensitive mat (xsensor, LX100:100.160.05, XSENSOR Technology Corporation, Calgary, Canada) | baseline
  Quantification of contact are between the patient and the mattress surface.
Contact area resulting from the exposure of patients to the supportive structures as detected by a pressure sensitive mat (xsensor, LX100:100.160.05, XSENSOR Technology Corporation, Calgary, Canada) | after 60 minutes of exposure to the mattress
  Quantification of contact are between the patient and the mattress surfaces.
Difference in stress assessment by means of heart rate | baseline
  Measurement of heart rate obtained from clinical routine patient surveillance.
Stress assessment by means of heart rate | after 60 minutes of exposure to the mattress
  Measurement of heart rate obtained from clinical routine patient surveillance.
Stress assessment by means of respiratory rate | baseline
  Measurement of respiratory rate obtained from clinical routine patient surveillance.
Stress assessment by means of respiratory rate | after 60 minutes of exposure to the mattress
  Measurement of respiratory rate obtained from clinical routine patient surveillance.
Stress assessment by means of blood pressure (mean arterial pressure) | baseline
  Measurement of blood pressure obtained from clinical routine patient surveillance.
Stress assessment by means of blood pressure (mean arterial pressure) | after 60 minutes of exposure to the mattress
  Measurement of blood pressure obtained from clinical routine patient surveillance.
Stress assessment by means of blood oxygen saturation | baseline
  Measurement of blood oxygen saturation obtained from clinical routine patient surveillance.
Stress assessment by means of blood oxygen saturation | after 60 minutes of exposure to the mattress
  Measurement of blood oxygen saturation obtained from clinical routine patient surveillance.
Stress assessment by means of body temperature | baseline
  Measurement of body temperature obtained from clinical routine patient surveillance.
Stress assessment by means of body temperature | after 60 minutes of exposure to the mattress
  Measurement of body temperature obtained from clinical routine patient surveillance.
Comfort assessment by means of a visual analogue scale | baseline
  Quantification of comfort level ranging from 0 [very uncomfortable] to 10 [very comfortable].
Comfort assessment by means of a visual analogue scale | after 60 minutes of exposure to the mattress
  Quantification of comfort level ranging from 0 [very uncomfortable] to 10 [very comfortable].
Stress assessment by means of a visual analogue scale | baseline
  Quantification of stress level ranging from 0 [totally relaxed] to 10 [very stressed].
Stress assessment by means of a visual analogue scale | after 60 minutes of exposure to the mattress
  Quantification of stress level ranging from 0 [totally relaxed] to 10 [very stressed].
Pain assessment by means of the questionnaire "Bern pain score for newborns - Revised (BSN-R)" | baseline
  Assessment of pain indicators (crying, facial expression, body tension, heart rate) ranging from 0 points (no pain indication) to 3 points (high pain indication). Total values >5 points for premature babies and >3 points for term babies is indicative for pain.
Pain assessment by means of the questionnaire "Bern pain score for newborns - Revised (BSN-R)" | after 60 minutes of exposure to the mattress
  Assessment of pain indicators (crying, facial expression, body tension, heart rate) ranging from 0 points (no pain indication) to 3 points (high pain indication). Total values >5 points for premature babies and >3 points for term babies is indicative for pain.
Unrest assessment by means of the Richmond Agitation-Sedation Scale (RASS) questionnaire | baseline
  Values range from -1 (sleepy) to 0 (attentive and calm) to +4 (belligerent).
Unrest assessment by means of the Richmond Agitation-Sedation Scale (RASS) questionnaire | after 60 minutes of exposure to the mattress
  Values range from -1 (sleepy) to 0 (attentive and calm) to +4 (belligerent).
Skin perfusion assessment by means of capillary refill time | baseline
  Assessment of the capillary refill time according to Jevon and Gallier (2020).
Skin perfusion assessment by means of capillary refill time | after 60 minutes of exposure to the mattress
  Assessment of the capillary refill time according to Jevon and Gallier (2020).
Skin assessment according to standard clinical procedure | baseline
  Identification and localisation (nose, mouth, occipital, face, ear, back, leg, foot, heel, others) of skin irregularities and evaluation of severity of irregularity (redness, partial injury of skin layers, all skin layers affected, complete tissue loss) according to clinical routine
Skin assessment by means of questionnaire | after 60 minutes of exposure to the mattress
  Identification and localisation (nose, mouth, occipital, face, ear, back, leg, foot, heel, others) of skin irregularities and evaluation of severity of irregularity (redness, partial injury of skin layers, all skin layers affected, complete tissue loss) according to clinical routine
Delirium assessment by means of the Cornell Assessment of Pediatric Delirium score (CAPD) | baseline
  Assessment of delirium indicators (eye contact, purposeful actions, awareness of surroundings, communication of needs, restlessness, refusal to be comforted, hypoactivity, response time) ranging from 0 points (not indicative for delirium) to 4 points (highly indicative for delirium). A delirium state is considered from a total value of >8 points.
Delirium assessment by means of the Cornell Assessment of Pediatric Delirium score (CAPD) | after 60 minutes of exposure to the mattress
  Assessment of delirium indicators (eye contact, purposeful actions, awareness of surroundings, communication of needs, restlessness, refusal to be comforted, hypoactivity, response time) ranging from 0 points (not indicative for delirium) to 4 points (highly indicative for delirium). A delirium state is considered from a total value of >8 points.
Withdrawal assessment by means of the Sophia Observation Withdrawal Symptoms scale (SOS) | baseline
  Assessment of withdrawal indicators (autonomic dysfunction [4 aspects], overstimulation of the central nervous system [9 aspects], dysfunction of the gastrointestinal tract [2 aspects] ranging from 0 points (not detectable) to 1 point (detectable). A withdrawal state is considered from a total value of >3 points.
Withdrawal assessment by means of the Sophia Observation Withdrawal Symptoms scale (SOS) | after 60 minutes of exposure to the mattress
  Assessment of withdrawal indicators (autonomic dysfunction [4 aspects], overstimulation of the central nervous system [9 aspects], dysfunction of the gastrointestinal tract [2 aspects] ranging from 0 points (not detectable) to 1 point (detectable). A withdrawal state is considered from a total value of >3 points.

CONTACTS AND LOCATIONS:
Overall Officials: Barbara Brotschi, Prof, Principal Investigator — Universitäts-Kinderspital Zürich, Zurich
Locations (1):
- University Children's Hospital Zurich, Zurich, Canton of Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: Yes
It is intended to publish the study in an open-access journal by December 2024. With this, the raw data of the interface pressure and contact area measurements will be made available upon request and fulfilling the access criteria as indicated below.
Supporting Information: Study Protocol, SAP
Time Frame: Data as indicated in the plan description will be available upon publication of the data Data will be available for an unlimited period of time.
Access Criteria: Data will be made available upon request for scientific analysis of the data. Research objectives and data analysis plan needs to be provided.

REFERENCES:
- [Background] Jevon P, Gallier H. How to measure capillary refill time in patients who are acutely ill. Nursing Times [online]. 2020; 116(8): 29-30.